CLINICAL TRIAL: NCT03963258
Title: Short-Term Effects of Whole-Body Vibration on Upper Extremity Function in Subjects With Poststroke Hemiplegia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Mouwang Zhou, Director, Head of Rehabilitation Medicine , Principal Investigator, Clinical Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00006761-M2018112
Record Dates: First submitted 2018-12-04; First posted 2019-05-24 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-07

CONDITIONS: Rehabilitation; Stroke; Hemiplegia; Physical Therapy Modalities; Electromyography; Upper Extremity; Recovery of Function; Vibration
Keywords: Whole-Body vibration; Stroke; Hemiplegia; upper extremity; Rehabilitation training; Muscular surface EMG; Vibration training
MeSH Terms: conditions — Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (Active Comparator): Over a 3-week period, the subjects in the control group received 1 hour daily of conventional upper limb training 5 times a week,including compensatory techniques for activities of daily living, UE strength, therapist-guided techniques for facilitating normal UE movement patterns,and range of motion and traditional positioning
  Interventions: Other: conventional upper limb training
- whole-body vibration group (Experimental): Subjects in the whole-body vibration group received half an hour of daily conventional upper limb training, followed by whole-body vibration training for an additional half hour per day,5 days per week during a 3-week period
  Interventions: Device: whole-body vibration training

INTERVENTIONS:
Device: whole-body vibration training — The subjects were exposed to alternating vertical sinusoidal vibration using a Galileo tilting table system.The frequency of WBV ranged from 5 to 20 Hz, and the amplitude ranged from 1 to 6 mm.The subjects were kneeled on the ground, both shoulders flexed at 90 degrees, elbows slightly flexed, their trunk bent in this position and contacted on the platform board with their palms equidistant from the midpoint of the board
  Other Names: vibration training
  Arms: whole-body vibration group
Other: conventional upper limb training — compensatory techniques for activities of daily living, UE strength, therapist-guided techniques for facilitating normal UE movement patterns,and range of motion and traditional positioning
  Arms: control group

SUMMARY:
To investigate the effect of whole body vibration on upper limb motor function in hemiplegic patients with subacute stroke

ELIGIBILITY:
Inclusion Criteria:

* After unilateral stroke 1 to 6 months
* An ischemic or hemorrhagic poststroke hemiplegia
* No cognitive impairment
* Able to reach Brunnstrom stage II or above in the proximal and distal parts of the arms
* No excessive pain in the more affected upper extremity
* All subjects agreed to participate in the study after receiving explanations regarding the purpose and procedures of the experiment, and they signed an informed consent statement before participation

Exclusion Criteria:

* Unsteadiness
* Accompanied by important organs (such as heart, liver, lung, kidney) dysfunction or malignant tumors
* Contraindications to general vibration training exist
* Combined with other diseases causing upper limb dysfunction

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-06-15 (Actual); Primary Completion 2020-05 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
upper-extremity Fugl-Meyer Scale | After the 3-week intervention period
  the assessment is scored by summing item ratings and reporting the aggregate score out of 66 points,with higher scores representing a greater UE motor ability summing item ratings and reporting the aggregate score out of 66 points, with higher scores representing a greater UE motor ability
Wolf Motor Function Test | After the 3-week intervention period
  participants were timed as they completed 15 activities that progressively involved more difficult arm movements and interactions with objects such as lifting a soda can, stacking checkers, and folding a towel. We reported the average time to perform the 15 items and the evaluator rated the normalcy of these items with a 6-point ordinal scale (range,0-5) using the functional ability scale.
Surface electromyography | After the 3-week intervention period
  Surface electromyography was used to measure the integrated EMG（IEMG）of the biceps and triceps during maximum isometric voluntary contraction（MIVC）of the affected elbow flexion and extension and then the co-contraction rate（CR）was calculated

CONTACTS AND LOCATIONS:
Overall Officials: mouwang zhou, master, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking Univercity Third Hospital, Beijing, No State Or Province, China

IPD SHARING:
Plan to Share IPD: Undecided